CLINICAL TRIAL: NCT07393126
Title: Effects of the Consumption of Test Product on Urination in Healthy Japanese Adults: A Randomized, Placebo-Controlled, Double-Blind, Parallel-Group Comparison Trial
Brief Title: Effects of the Consumption of Test Product on Urination in Healthy Japanese Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indena S.p.A (Industry)
Collaborators: Orthomedico Inc. (Other); Indena Japan Co. LTD (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 01170-0018-29; UMIN000060011 (Registry Identifier: UMIN-CTR)
Record Dates: First submitted 2026-01-21; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Healthy Japanese
Keywords: Cranberry; Urination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cranberry Phospholipids (Active Comparator): Take two tablets (containing 120 mg cranberry phospholipids/tablet)
  Interventions: Dietary Supplement: Cranberry Phospholipids
- Placebo (Placebo Comparator): Take two tablets (containing 0 mg cranberry phospholipids/tablet)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Cranberry Phospholipids — Take two tablets will be taken once daily
  Arms: Cranberry Phospholipids
Dietary Supplement: Placebo — Take two tablets will be taken once daily
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to test in Japanese adults who experience concerns regarding urinary frequency. The main question it aims to answer is:

•Does consumption of Cranberry Phospholipids reduce daytime urinary frequency?

Participants will be given the following tasks:

* Take two tablets daily containing Cranberry Phospholipid for eight weeks.
* Answer the questionnaire on the overactive bladder (OAB)-specific quality of life (QOL).
* Answer the questionnaire on OAB symptoms.
* Answer the questionnaire on urinary frequency during the study period. Researchers will compare Cranberry Phospholipids and placebo groups to see if Cranberry Phospholipids reduces daytime urinary frequency.

ELIGIBILITY:
Inclusion Criteria:

* Japanese
* Men or women
* Adults
* Healthy individuals
* Individuals with positive urine leukocytes at baseline
* Individuals whose score of urinary urgency of overactive bladder symptom score (OABSS) is less than two or total score of OABSS is less than three at baseline
* Individuals whose "frequent urination during the daytime hours" of "symptom bother" of OAB-q is relatively high at baseline

Exclusion Criteria:

* Individuals undergoing medical treatment or having a medical history of malignant tumor, heart failure, or myocardial infarction
* Individuals carrying a pacemaker or an implantable cardioverter defibrillator
* Individuals undergoing treatment for any of the following chronic diseases: cardiac arrhythmia, liver disease, kidney disease, cerebrovascular disorder, rheumatism, diabetes mellitus, dyslipidemia, hypertension, or any other chronic diseases
* Individuals who use or take "Foods for Specified Health Uses", "Foods with Functional Claims", or other functional food/beverage as part of their daily diet
* Individuals currently regularly taking medications (including herbal medicines) and supplements
* Individuals who are allergic to medicines and/or the test-product-related products in this trial
* Individuals with urinary pain
* Individuals undergoing treatment, have had treatment within two months, or need the treatment for diseases related to urination, e.g. benign prostatic hypertrophy, prostatitis, prostate cancer, overactive bladder, hypoactive bladder, cystitis, interstitial cystitis, bladder cancer, bladder stones, urethritis, urethral stricture, neurological disease, polyuria, and nocturnal polyuria
* Individuals have overactive bladder symptom (individuals who urinate eight times or more per day, and have urinary urgency at least once a week)
* Individuals wake up twice or more to urinate at bedtime
* Individuals are pregnant, breast-feeding, and planning to become pregnant
* Individuals have been enrolled in other clinical trials within the last 28 days before the agreement to participate in this trial or plan to participate another trial during this trial
* Individuals are judged as ineligible to participate in the trial by the physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-12-08 (Actual); Primary Completion 2026-06-19 (Estimated); Study Completion 2026-06-19 (Estimated)

PRIMARY OUTCOMES:
Measured value for the Overactive Bladder Questionnaire (OAB-q) questionnaire item "frequent urination during the daytime hours" after the 8-week intervention | After the 8-week intervention
  Using OAB-q, we evaluate OAB-specific quality of life (QOL). The questionnaire have 33 items, including 8 items measuring "symptom bother" and 25 items measuring "impact on QOL," with each item rated on a 6-point scale."Impact on QOL" is scored across four domains: "Coping" (8 items), "Concern" (7 items), "Sleep" (5 items), and "Social Interaction" (5 items). Scores are calculated on a scale of 0 to 100, with higher scores indicating a greater degree of difficulty. On the other hand, the "impact on QOL" indicates that the higher the score, the better the QOL.

SECONDARY OUTCOMES:
Individuals whose the response to the OAB-q questionnaire item "frequent urination during the daytime hours" improved by one or more scale points after the 8-week intervention compared to Baseline | Baseline, and after the 8-week intervention
  Using OAB-q, we evaluate OAB-specific QOL. The questionnaire have 33 items, including 8 items measuring "symptom bother" and 25 items measuring "impact on QOL," with each item rated on a 6-point scale."Impact on QOL" is scored across four domains: "Coping" (8 items), "Concern" (7 items), "Sleep" (5 items), and "Social Interaction" (5 items). Scores are calculated on a scale of 0 to 100, with higher scores indicating a greater degree of difficulty. On the other hand, the "impact on QOL" indicates that the higher the score, the better the QOL.
The amount of change, and percentage of change from Baseline for the OAB-q questionnaire item "frequent urination during the daytime hours" after the 8-week intervention | Baseline, after the 1-week intervention, the 3-week intervention and the 8-week intervention
  Using OAB-q, we evaluate OAB-specific QOL. The questionnaire have 33 items, including 8 items measuring "symptom bother" and 25 items measuring "impact on QOL," with each item rated on a 6-point scale."Impact on QOL" is scored across four domains: "Coping" (8 items), "Concern" (7 items), "Sleep" (5 items), and "Social Interaction" (5 items). Scores are calculated on a scale of 0 to 100, with higher scores indicating a greater degree of difficulty. On the other hand, the "impact on QOL" indicates that the higher the score, the better the QOL.
The measured values, amount of changes, and percentage of changes from Baseline for all other questionnaire items of the OAB-q, excluding "frequent urination during the daytime hours," after the 8-week intervention | Baseline, after the 1-week intervention, the 3-week intervention and the 8-week intervention
  Using OAB-q, we evaluate OAB-specific QOL. The questionnaire have 33 items, including 8 items measuring "symptom bother" and 25 items measuring "impact on QOL," with each item rated on a 6-point scale."Impact on QOL" is scored across four domains: "Coping" (8 items), "Concern" (7 items), "Sleep" (5 items), and "Social Interaction" (5 items). Scores are calculated on a scale of 0 to 100, with higher scores indicating a greater degree of difficulty. On the other hand, the "impact on QOL" indicates that the higher the score, the better the QOL.
The measured values, and amount of changes and percentage of changes from Period 1 for the average frequency of urination during the daytime, during the nighttime, and all day, as measured during Periods 2 to 9 | Period 1 (7 days prior to Baseline), Period 2~9 (periods separated by 7 days from the start of intervention)
  Participants will maintain a daily diary of their urination frequency during two distinct periods: for 7 days immediately preceding the Baseline, and from the beginning of the intervention until the day before the final examination.
Individuals who experienced adverse events | After the 8-week intervention
  During the trial period, if a participant exhibits any clinically significant "new manifestation of abnormality" or "aggravation" in his/her physical signs and symptoms, it is considered to be an adverse event.
Individuals whose values of urinalysis and peripheral blood test are outside the reference range after intervention despite within the reference range at Baseline | Baseline, and after the 8-week intervention
  The ratio of cases which had test items stated in urinalysis and peripheral blood examination within their respective standard ranges before intervention but exceeded the ranges after intervention are calculated, intergroup comparison at each time point is performed using tests for comparing proportions.
Body height | Baseline, and after the 8-week intervention
  Body height is measured using a height meter.
Body weight | Baseline, and after the 8-week intervention
  Body weight is measured using a body scale.
Blood pressure | Baseline, and after the 8-week intervention
  Systolic and diastolic blood pressure are measured using a digital wrist-type sphygmomanometer.
Urinalysis | Baseline, and after the 8-week intervention
  A urine sample (approximately 10 mL) will be collected from each participant, and the samples will be sent to LSI Medience Corporation for analysis.
Peripheral blood examination | Baseline, and after the 8-week intervention
  A venous blood sample (approximately 10 mL) will be collected from each participant, and the samples will be sent to LSI Medience Corporation for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Tsuyoshi Takara, MD, Study Chair — Medical Corporation Seishinkai, Takara Clinic
Locations (2):
- Japan (2):
  - Nerima Medical Association Minami-machi Clinic, Nerima-ku, Tokyo
  - Medical Corporation Seishinkai, Takara Clinic, Shinagawa-Ku, Tokyo

IPD SHARING:
Plan to Share IPD: No
Data sharing will be discussed among the research affiliates after the study is completed.